CLINICAL TRIAL: NCT01914796
Title: A Phase 1, Double Blind, Sponsor Open, Randomized, Placebo Controlled, Crossover, Single Oral Dose Escalation Study To Investigate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-06412562 In Healthy Subjects
Brief Title: A Phase I Trial to Investigate the Safety and Tolerability of PF-06412562
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B7441001
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Phase 1; Randomized; Double Blind; Placebo-Controlled; Single-Dose Escalation; Safety; Tolerability; PK; PD; PF-06412562

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single ascending doses (Placebo Comparator)
  Interventions: Drug: PF-06412562
- Measurement of eye blink rate (Placebo Comparator)
  Interventions: Drug: PF-06412562

INTERVENTIONS:
Drug: PF-06412562 — Single doses, given by oral solution, starting at 0.5 mg up to a possible maximum of 150 mg. The subject will have been fasted for 10 hours prior to the single dose. Two doses, 120 mg and 150 mg, will be split into 3 doses such that the total dose is given over 8 hours (i.e. t = 0, 4, and 8 hours). For each dosing period, 2 subjects will be given a placebo as a comparator. One dose will be given in the fed state.
  Arms: Single ascending doses
Drug: PF-06412562 — It is believed that for increasing doses of this compound the eye blink rate (EBR) will also increase. This arm will use EBR measurement technology to verify this hypothesis. In each dosing period, 4 subjects will be given a placebo as a comparator.
  Arms: Measurement of eye blink rate

SUMMARY:
This study will determine the safety and tolerability of PF-06412562 given orally to healthy volunteers. To determine the optimal dose for future studies, the concentration of the drug over time will be determined by periodic blood samples. The rate of eye blinks will be measured as an indicator of PF-06412562 action on the receptors of interest in the brain.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years

Female subjects of non childbearing potential that meet at least one of the following criteria:

Achieved postmenopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal status;

* Have undergone a documented hysterectomy and/or bilateral oophorectomy;
* Have medically confirmed ovarian failure.

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Any condition possibly affecting drug absorption .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Plasma Decay Half-Life (t1/2) | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
  AUC = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time. It is obtained from AUC (0 - t) plus AUC (t - 8).
Apparent Oral Clearance (CL/F) | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24, 32 hours post-dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Measurement of Cognitive Decline by Means of a Computerized Battery of Neuropsychologic Tests | 0, 1, 4, 8, 12 hours post-dose
  Change from baseline cognitive performance
Eye Blink Rate | 0, 1, 2, 4 and 8 hours
  Measurement of eye blink rate for a given dose at time of predicted maximum blood concentration of the compound.
Area Under the Curve From Time Zero to 24 hours | 0, 0.5, 1, 1.5, 2, 4, 5, 6, 8, 9, 10, 12, 16, 24 hours post-dose
  Area under the plasma concentration time-curve from zero to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441001&StudyName=A%20Phase%20I%20Trial%20to%20Investigate%20the%20Safety%20and%20Tolerability%20of%20PF-06412562